CLINICAL TRIAL: NCT06502574
Title: Strengthening Participation in Social Life Through Rational Drug Use and Disease Self-Care Management inOlder Adults
Brief Title: Self-Care Management in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Ayaz Alkaya (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor-Investigator, Sultan Ayaz Alkaya, Prof. Dr., Faculty of Nursing, Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-341
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Disease Self Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile application (Experimental): Older adults will be asked to use the mobile application for atleast 6 months, and the scales will be re-administered face toface or online in the 3rd and 6th months of the intervention.
  Interventions: Other: mobile application
- Control (No Intervention): No intervention has been made.

INTERVENTIONS:
Other: mobile application — The mobile application prepared for rational drug use andchronic disease self-management, suitable for use by olderadults, will be required to be used for 6 months.
  Arms: mobile application

SUMMARY:
Self-management of chronic diseases requires the ability to manage the symptoms, treatment, and lifestyle changes inherent in living with achronic disease. Rational drug use by older adults is of particular importance. Mobile applications are being developed to facilitate thecompliance of older adults with chronic diseases with medication treatment and to increase their disease self-management skills. The researchwas planned to strengthen participation in social life through rational drug use and disease self-care management in older adults with chronicdiseases. The research will be conducted in a parallel group randomized controlled manner. In the research, a mobile application will bedeveloped for the use of older adults. Older adults will be asked to use the mobile application for at least 6 months, and the scales will be re-administered face to face or online in the 3rd and 6th months of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 60-79 age group,
* Having a chronic disease that requires constant monitoring and treatment
* Using at least one medication for your disease regularly
* Having smart phone usage skills

Exclusion Criteria:

* Having vision and hearing problems
* Being 80 or older
* Having a neuro-psychiatric disease

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Participation in social life (Social Inclusion Scale) | Baseline
  It was developed in 2009 by Secker et al. to measure an individual's relationship with other people. A validity and reliability study of theTurkish version of the scale was conducted. 4 items were removed from the original 22-item scale and the final version consisted of 18items. The lowest and highest that can be taken from the scale are 18 and 72. A higher score from the scale indicates more socialization.
Participation in social life (Social Inclusion Scale) | within first week]
  It was developed in 2009 by Secker et al. to measure an individual's relationship with other people. A validity and reliability study of theTurkish version of the scale was conducted. 4 items were removed from the original 22-item scale and the final version consisted of 18items. The lowest and highest that can be taken from the scale are 18 and 72. A higher score from the scale indicates more socialization.
Participation in social life (Social Inclusion Scale) | twelfth week]
  It was developed in 2009 by Secker et al. to measure an individual's relationship with other people. A validity and reliability study of theTurkish version of the scale was conducted. 4 items were removed from the original 22-item scale and the final version consisted of 18items. The lowest and highest that can be taken from the scale are 18 and 72. A higher score from the scale indicates more socialization.